CLINICAL TRIAL: NCT00005258
Title: Family Study of Congenital Cardiovascular Malformations
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1141; R01HL044069 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2001-11

CONDITIONS: Cardiovascular Diseases; Defect, Congenital Heart; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Defects, Congenital; Heart Diseases

SUMMARY:
To determine genetic mechanisms responsible for congenital cardiovascular malformations.

DETAILED DESCRIPTION:
BACKGROUND:

Congenital cardiovascular malformations are a major cause of infant mortality in the United States. In 1985, six defects -- hypoplastic left heart, tetralogy of Fallot, truncus arteriosus, transposition of the great arteries, endocardial cushion defect, and ventricular septal defect -- were among the fifteen most frequent causes of premature death due to congenital malformations, accounting for 109,063 years of life lost. This loss of productive life continues in spite of major advances in medical and surgical treatment of congenital cardiovascular malformations. Even as successful treatment modalities are developed, the survival to reproductive years without improved understanding of genetic risks produces additional unanswered questions.

DESIGN NARRATIVE:

Clinical assessment of cases and controls included medical history, pedigree construction, complete evaluation by a pediatric cardiologist, and two-dimensional and Doppler echocardiography. First degree relatives of cases and controls underwent clinical-echocardiographic evaluation also. The distribution of cardiac defects for all pedigrees within and among the proband group was delineated. The frequencies of heart defects were compared within and among pedigrees of cases and controls. Regressive logistic models of genetic determinants for the malformations were tested. The three participating clinical centers included University of Maryland at Baltimore, the Johns Hopkins Hospital, and the University of Rochester in Rochester, New York.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-06; Study Completion 1993-05 (Actual)